CLINICAL TRIAL: NCT01019928
Title: A Phase IIa, Double-blind, Randomized, 2-way Cross-over Study to Evaluate the Effect of a Single Dose of AZD1386 95 mg Compared to Placebo in a Multimodal Experimental Pain Model on Esophageal Sensitivity in GERD Patients With a Partial Response to PPI Treatment
Brief Title: Esophageal Hypersensitivity Study in Patients With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D9127C00002; 2008-007420-26
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-10

CONDITIONS: Sensitivity in Esophagus
Keywords: GERD; patient; esophagus; pain
MeSH Terms: conditions — Gastroesophageal Reflux; Pain | interventions — AZD1386

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- First AZD1386, then washout, then placebo (Experimental)
  Interventions: Drug: AZD1386; Drug: Placebo to AZD1386
- First placebo, then washout, then AZD1386 (Experimental)
  Interventions: Drug: AZD1386; Drug: Placebo to AZD1386

INTERVENTIONS:
Drug: AZD1386 — 95 mg, oral solution, single dose
Drug: Placebo to AZD1386 — Placebo, oral solution, single dose

SUMMARY:
The purpose of the study is to compare sensitivity of visceral pain in the esophagus using different pain stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent form
* BMI 18.5-35.0, inclusive
* Continuous PPI treatment for GERD during the last 4 weeks

Exclusion Criteria:

* Patients that have not experienced any GERD symptoms improvement at all after PPI treatment
* Unstable or clinically significant disorders including cardiovascular, respiratory, renal, hepatic, metabolic, psychiatric, other gastrointestinal and esophageal disorders besides GERD
* Prior surgery of the upper GI tract

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Sundin, Study Director — AstraZeneca R&D, Mölndal, Sweden; Peter Funch-Jensen,, MD, PhD, Principal Investigator — Aarhus Hospital, Dept of Surgical Gastroenterology, Aarhus, Denmark
Locations (2):
- Research Site, Århus C, Denmark
- Research Site, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Krarup AL, Ny L, Gunnarsson J, Hvid-Jensen F, Zetterstrand S, Simren M, Funch-Jensen P, Hansen MB, Drewes AM. Randomized clinical trial: inhibition of the TRPV1 system in patients with nonerosive gastroesophageal reflux disease and a partial response to PPI treatment is not associated with analgesia to esophageal experimental pain. Scand J Gastroenterol. 2013 Mar;48(3):274-84. doi: 10.3109/00365521.2012.758769. Epub 2013 Jan 16. PMID 23320520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 patients were enrolled, 16 of these patients were NOT randomized for the following reasons:
  Voluntary discontinuation by patient = 3 Incorrect enrollment (did not meet inclusion/excl criteria) = 13
Pre-assignment Details: 14 patients were randomised, 1 patient received placebo in the first treatment period without any events, but had an SAE prior to receiving AZD1386 in the second period and was withdrawn. 13 randomised patients completed the study, but one of these patients was incorrectly enrolled and excluded from the per-protocol analysis set.
Period: Period 1
Arm/Group | First AZD1386, Then Washout, Then Placebo | First Placebo, Then Washout, Then AZD1386
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Period 2
Arm/Group | First AZD1386, Then Washout, Then Placebo | First Placebo, Then Washout, Then AZD1386
Started | 7 | 7
Completed | 7 | 6 (One patient had an SAE, and was withdrawn, prior to receiving AZD1386)
Not Completed | 0 | 1
Period: Period 3
Arm/Group | First AZD1386, Then Washout, Then Placebo | First Placebo, Then Washout, Then AZD1386
Started | 7 | 6 (One patient had an SAE, and was withdrawn, prior to receiving AZD1386)
Completed | 7 | 6 (One patient had an SAE, and was withdrawn, prior to receiving AZD1386)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1386 95 mg | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 54.9 (15.0) | 54.7 (17.4) | 54.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Visual Analogue Scale 7 (VAS7) During Thermal Stimulation at 1.5 Hours Post-Dose.
Description: A probe (bag) was inserted 7cm above the lower esophageal sphincter (LES). Heat stimuli were applied by recirculation of heated water in the bag. Prior to recirculation the bag is filled with 7mL to ensure adequate mucosal contact. Water was heated up to a maximum of 63° C and the stimulation was continued until VAS 7 was reached.
  The intensities of the non-painful sensations were scored with the following descriptors added to facilitate the scoring:
  1. = vague perception of mild sensation
  2. = definite perception of mild sensation
  3. = vague perception of moderate sensation
  4. = definite perception of moderate sensation
     For painful sensations the patients will use the scale from 5-10 anchored at:
  5. = pain detection
  6. = slight pain
  7. = moderate pain
  8. = medium pain intensity
  9. = intense pain
  10. = unbearable pain
Time Frame: 1.5 hours post dose
Measure: Geometric Mean (Full Range); unit: seconds
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 13
seconds | 84.0 [36 to 146] | 86.9 [29 to 127]

2. Secondary Outcome: Time to Visual Analogue Scale 7 (VAS7) During Thermal Stimulation at 0.5 Hours Post Dose
Description: as for outcome 1
Time Frame: 0.5 hours post dose
Measure: Geometric Mean (Full Range); unit: seconds
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 13
seconds | 86.0 [41 to 157] | 87.8 [31 to 132]

3. Secondary Outcome: Time to Visual Analogue Scale 7 (VAS7) During Thermal Stimulation at 2.5 Hours Post Dose
Description: as for outcome 1
Time Frame: 2.5 hours post dose
Measure: Geometric Mean (Full Range); unit: seconds
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 13
seconds | 85.5 [39 to 150] | 77.0 [24 to 125]

4. Secondary Outcome: Volume at Visual Analogue Scale 7 (VAS7) During Mechanical Stimulation at 0.5 Hours Post Dose
Description: A probe (bag) was inserted 7cm above the lower esophageal sphincter (LES). Volume change in the bag was recorded continuously at each level of the visual analogue scale (VAS) and up to VAS7 (Volume at Visual Analogue Scale 7).
  The intensities of the non-painful sensations were scored with the following descriptors added to facilitate the scoring:
  1. = vague perception of mild sensation
  2. = definite perception of mild sensation
  3. = vague perception of moderate sensation
  4. = definite perception of moderate sensation
     For painful sensations the patients will use the scale from 5-10 anchored at:
  5. = pain detection
  6. = slight pain
  7. = moderate pain
  8. = medium pain intensity
  9. = intense pain
  10. = unbearable pain
Time Frame: 0.5 hours post dose
Measure: Geometric Mean (Full Range); unit: ml
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 13
ml | 16.2 [8 to 37] | 15.1 [6 to 41]

5. Secondary Outcome: Volume at Visual Analogue Scale 7 (VAS7) During Mechanical Stimulation at 1.5 Hours Post-Dose
Description: as for outcome 4
Time Frame: 1.5 hours post dose
Measure: Geometric Mean (Full Range); unit: ml
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 13
ml | 15.0 [8 to 24] | 16.7 [8 to 30]

6. Secondary Outcome: Volume at Visual Analogue Scale 7 (VAS7) During Mechanical Stimulation at 2.5 Hours Post-Dose.
Description: as for outcome 4
Time Frame: 2.5 hours post dose
Measure: Geometric Mean (Full Range); unit: ml
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 11 | 13
ml | 15.4 [6 to 29] | 15.2 [5 to 38]

7. Secondary Outcome: Current at Visual Analogue Scale 7 (VAS7) During Electrical Stimulation 0.5 Hours Post Dose
Description: A probe (bag) was inserted 7cm above the lower esophageal sphincter (LES) and stimulations were performed at approximately 8 cm above the LES. The intensity of the stimuli is increased steadily in steps of 0.5 to 1 mA and the intensity corresponding to the VAS levels 1, 3, 5 and 7 were recorded.
  The current will be increased until the patient report moderate pain (VAS 7) or max 80 mA.
  The intensities of the non-painful sensations were scored with the following descriptors added to facilitate the scoring:
  1. = vague perception of mild sensation
  2. = definite perception of mild sensation
  3. = vague perception of moderate sensation
  4. = definite perception of moderate sensation
     For painful sensations the patients will use the scale from 5-10 anchored at:
  5. = pain detection
  6. = slight pain
  7. = moderate pain
  8. = medium pain intensity
  9. = intense pain
  10. = unbearable pain
Time Frame: 0.5 hours post dose
Measure: Geometric Mean (Full Range); unit: mA
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 12
mA | 16.7 [9 to 31] | 16.7 [9 to 40]

8. Secondary Outcome: Current at Visual Analogue Scale 7 (VAS7) During Electrical Stimulation at 1.5 Hours Post Dose
Description: as for outcome 7
Time Frame: 1.5 hours post dose
Measure: Geometric Mean (Full Range); unit: mA
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 12
mA | 16.7 [8 to 30] | 15.8 [8 to 37]

9. Secondary Outcome: Current at Visual Analogue Scale 7 (VAS7) During Electrical Stimulation at 2.5 Hours Post Dose
Description: as for outcome 7
Time Frame: 2.5 hours post dose
Measure: Geometric Mean (Full Range); unit: mA
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 11 | 12
mA | 16.2 [8 to 31] | 14.8 [8 to 28]

10. Secondary Outcome: AUCt
Description: Area under the plasma concentration curve from time zero to the last quantifiable concentration
Time Frame: 0 to 4 hours post dose
Measure: Geometric Mean (95% Confidence Interval); unit: nmol*h/L
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 0
nmol*h/L | 5899 [4735 to 7349] |

11. Secondary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: 0 to 4 hours post dose
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 0
nmol/L | 2361 [1859 to 3000] |

12. Secondary Outcome: Tmax
Description: Time of maximum plasma concentration
Time Frame: 0 to 4 hours post dose
Measure: Median (Full Range); unit: hours
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 12 | 0
hours | 1.0 [0.5 to 2.5] |

13. Secondary Outcome: SBP
Description: Supine Systolic Blood Pressure at 1.5 hours post dose
Time Frame: 1.5 hours post dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 13 | 14
mmHg | 145.8 (10.3) | 139.7 (12.7)

14. Secondary Outcome: DBP
Description: Supine Diastolic Blood Pressure at 1.5 hours post dose
Time Frame: 1.5 hours post dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 13 | 14
mmHg | 81.4 (8.1) | 80.0 (7.3)

15. Secondary Outcome: Pulse
Description: Supine Pulse at 1.5 hours post dose
Time Frame: 1.5 hours post dose
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 13 | 14
beats/min | 67.8 (12.9) | 62.2 (9.4)

16. Secondary Outcome: QTcF
Description: QT interval corrected for heart rate using Fredericia formula(QTcF) at 1.5 hours post dose
Time Frame: 1.5 hours post dose
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 13 | 14
ms | 409.6 (19.0) | 414.3 (17.3)

17. Secondary Outcome: Body Temperature
Description: Oral Body Temperature at 1.5 hours post dose
Time Frame: 1.5 hours post dose
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 13 | 14
degrees Celsius | 37.2 (0.4) | 36.8 (0.3)

18. Secondary Outcome: Clinically Relevant Change of Laboratory Variables
Description: Number of participants with clinically relevant change of laboratory variables(clinical chemistry, haematology and urinalysis parameters)
Time Frame: Pre-entry to follow-up
Measure: Number; unit: Participants
Arm/Group | AZD1386 95 mg | Placebo
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | AZD1386 95 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/14
Other Adverse Events (participants affected / at risk) | 11/13 | 2/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1386 95 mg (N=13) | Placebo (N=14)
ECG, atrial fibrillation (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1386 95 mg (N=13) | Placebo (N=14)
Feeling Cold (General disorders) | 7 | 0
Chills (General disorders) | 1 | 0
Feeling Of Body Temperature Change (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Hypoaesthesia Oral (General disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal Disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Body Temperature Increased (Investigations) | 4 | 0
Ageusia (Nervous system disorders) | 1 | 0
Burning Sensation (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral Coldness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days